CLINICAL TRIAL: NCT06138483
Title: A New Mutational and Epigenetic Signature to Predict Early OPSCC Relapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO 2019.13
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inclusion of new biomarkers to improve the personalized treatment approach for HPV-positive and -negative oropharyngeal squamous cell carcinoma (OPSCC) patients is urgently needed. Emerging evidences suggest that mutations in epigenetic regulators, as well as epigenetic changes, deeply influence the biology of OPSCC, thus representing attractive targets for the definition of novel molecular markers for this malignancy. Based on these considerations, our project aims to retrospectively identify a new mutational and epigenetic signature to identify OPSCC patients at high risk of early relapse, and to set up a new multicenter prospective study in order to validate it

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed, previously untreated, histologically confirmed stage III-IVa OPSCC, according to AJCC 7th Edition,
* managed with definitive treatment modality (either radical surgery plus adjuvant radiotherapy ± chemotherapy or definitive chemo-radiotherapy)
* minimum follow up of 2 years or who had disease recurrence within 2 years after the end of treatment.
* neoplastic lesion contains ≥ 70% neoplastic cells

Exclusion Criteria:

Patients:

* with distant metastases at diagnosis,
* who have been managed with palliative intent;
* with previous history of head and neck cancer are not eligible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caucasian patients, with newly diagnosed, previously untreated, histologically confirmed stage III-IVa OPSCC
Sampling Method: Non-Probability Sample
Enrollment: 267 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
risk of recurrence | 18 months
  risk of recurrence in patients with a negative prognostic epigenetic signature compared to patients with a positive one

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Fratta, PhD, Principal Investigator — Centro di Riferimento Oncologico (CRO), IRCCS
Locations (5):
- Italy (5):
  - Centro di Riferimento Oncologico (CRO), IRCCS, Aviano
  - Ospedale San Martino di Belluno - ULSS 1 Dolomiti, Belluno
  - Ospedale dell'Angelo - Mestre - Ulss 3 Serenissima, Mestre
  - Ospedale Santa Maria degli Angeli - ASFO, Pordenone
  - Ospedale di Treviso - ULSS 2 Marca Trevigiana, Treviso

IPD SHARING:
Plan to Share IPD: No